CLINICAL TRIAL: NCT01197326
Title: The Use of IntelliVue Patient Monitor MP5 Rel. G.1 for the Prevention of "Failure to Rescue" Using Early Warning Score
Brief Title: The Prevention of Failure to Rescue Using Early Warning Scoring
Acronym: VitalCare
Status: Completed | Type: Observational
Sponsor: Philips Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: BUD33108
Record Dates: First submitted 2010-09-03; First posted 2010-09-09 (Estimated); Results first posted 2014-11-20 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-04

CONDITIONS: Sepsis; Renal Failure; Pulmonary Edema; Cardio-pulmonary Arrest
Keywords: patient deterioration; unplanned ICU admissions; rapid response teams
MeSH Terms: conditions — Sepsis; Renal Insufficiency; Pulmonary Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: Patients who triggered MET/RRT calls prior to the use of the MP5 EWS patient monitor.
  Interventions: Device: use of the MP5 EWS patient monitor
- Group 2: Patients who triggered MET/RRT calls after the use of the MP5 EWS patient monitor.
  Interventions: Device: use of the MP5 EWS patient monitor

INTERVENTIONS:
Device: use of the MP5 EWS patient monitor — All patients on the study ward receive the same care in Groups 1 and 2. The only difference is the device used to collect the vital signs. In Group 2, the MP5 EWS spot check monitor (FDA approved and CE marked) is the vital signs collection device.

SUMMARY:
The purpose of this study is to assess if, compared with standard paper-based systems, an automated Early Warning System (EWS) resident in a spot check patient monitor, can help to identify deteriorating patients.

DETAILED DESCRIPTION:
The purpose of this study is to assess if, compared with standard paper-based systems, an automated Early Warning System (EWS) resident in a spot check patient monitor, can help to identify patients in the acute care settings but outside of the intensive care unit, who may be experiencing physiological instability and who are in need of rapid clinical intervention by a Rapid Response Team (RRT)/ Medical Emergency Team (MET).

The development of such an automated system by offers a unique opportunity to assess its user-friendliness, labour-saving effect, feasibility and clinical utility. Accordingly, we plan to conduct a research program aimed at assessing this new approach toward patient monitoring.

This study will use the hospital's Standard of Care protocol for the monitoring of vital signs (including timing and vital signs collected) and a commercially available automatic spot check monitor to collect data. No investigational procedures or devices are associated with this protocol.

ELIGIBILITY:
Inclusion Criteria:

* all patients admitted to the study units during the period of data collection

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We plan to observe a non-probability, convenience sample of patients which will consist primarily of acutely ill hospitalized adult patients (at least 18 years of age). We will also enroll 1-2 pediatric units to be used as pilot data, since there is less available empiric data published in the literature. Study participants will be recruited from all eligible patients during the enrollment period who are having vital signs monitoring performed as Standard of Care.
Sampling Method: Non-Probability Sample
Enrollment: 414 (Actual)
Dates: Start 2009-08; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rinaldo Bellomo, MD, Principal Investigator — Faculty of Medicine, University of Melbourne, Melbourne, Australia
Locations (1):
- Austin Hospital, Heidelberg, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bellomo R, Ackerman M, Bailey M, Beale R, Clancy G, Danesh V, Hvarfner A, Jimenez E, Konrad D, Lecardo M, Pattee KS, Ritchie J, Sherman K, Tangkau P; Vital Signs to Identify, Target, and Assess Level of Care Study (VITAL Care Study) Investigators. A controlled trial of electronic automated advisory vital signs monitoring in general hospital wards. Crit Care Med. 2012 Aug;40(8):2349-61. doi: 10.1097/CCM.0b013e318255d9a0. PMID 22809908

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 439 beds in 12 general wards in 10 hospital from five countries inthe USA, Europe and Australia.
Groups:
- Group 1: Patients who triggered MET/RRT calls prior to the use of the MP5 EWS patient monitor.
  Use the MP5 EWS monitor to measure routine vital signs : All patients on the study ward receive the same care in Groups 1 and 2. The only difference is the device used to collect the vital signs. In Group 2, the MP5 EWS spot check monitor (FDA approved and CE marked) is the vital signs collection device.
- Group 2: Patients who triggered MET/RRT calls after the use of the MP5 EWS patient monitor.
  Use the MP5 EWS monitor to measure routine vital signs : All patients on the study ward receive the same care in Groups 1 and 2. The only difference is the device used to collect the vital signs. In Group 2, the MP5 EWS spot check monitor (FDA approved and CE marked) is the vital signs collection device.
Period: Overall Study
Arm/Group | Group 1 | Group 2
Started | 205 | 209
Completed | 205 | 209
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 205 | 209 | 414
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 82 | 73 | 155
  >=65 years | 123 | 136 | 259
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (13.2) | 70.1 (15.6) | 69.3 (15.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 103 | 202
  Male | 106 | 106 | 212
Region of Enrollment [Number; unit: participants]
  Australia | 42 | 38 | 80
  United States | 124 | 118 | 242
  Sweden | 21 | 20 | 41
  Netherlands | 7 | 9 | 16
  United Kingdom | 11 | 24 | 35

OUTCOME MEASURES:

1. Primary Outcome: Survival
Description: Survival at the end of the RRT call (time when the RRT team left the patient, average duration of calls around 25 min)
Time Frame: 6 months
Measure: Number; unit: percentage of participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 205 | 209
percentage of participants | 86 | 92

2. Secondary Outcome: Respiration Rate Impact on RRT Calls
Description: Proportion of calls secondary to abnormal respiratory vital signs. Respiration Rate is considered to be one of the main early indicators of deterioration.
Time Frame: 6 months
Measure: Number; unit: percentage of calls
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 205 | 209
percentage of calls | 21 | 31

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Patients Who Triggered MET/RRT Calls Prior to the Use of MP5: Patients who triggered MET/RRT calls prior to the use of the MP5 EWS patient monitor
- Patients Who Triggered MET/RRT Calls After the Use of MP5: Patients who triggered MET/RRT calls after the use of the MP5 EWS patient monitor
Arm/Group | Patients Who Triggered MET/RRT Calls Prior to the Use of MP5 | Patients Who Triggered MET/RRT Calls After the Use of MP5
Serious Adverse Events (participants affected / at risk) | 0/205 | 0/209
Other Adverse Events (participants affected / at risk) | 0/205 | 0/209

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less